CLINICAL TRIAL: NCT06366919
Title: Comparison of Effectiveness of Alexander Technique Versus Feldenkrais Technique in Non - Specific Neck Pain Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DPT/Batch-Fall19/559
Record Dates: First submitted 2024-04-03; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alexander Technique (AT) (Experimental)
  Interventions: Diagnostic Test: Alexander Technique (AT)
- Feldenkrais Technique (FT) (Experimental)
  Interventions: Diagnostic Test: Feldenkrais Technique (FT)

INTERVENTIONS:
Diagnostic Test: Alexander Technique (AT) — The AT arm of study will involve participants receiving indivisual sessions. These sessions will typically focus on non specific neck pain management improving posture , movement coordination and body awareness through gentle hands on guidance
  Arms: Alexander Technique (AT)
Diagnostic Test: Feldenkrais Technique (FT) — The FT arm of study will involve participants recieving individual sessions. These sessions will typically focus on pain improvement, maintaining alignment, reducing muscle tension and promoting ease of movement.
  Arms: Feldenkrais Technique (FT)

SUMMARY:
Comparison of Effectiveness of Alexander Technique Versus Feldenkrais Technique in Non - Specific Neck Pain Patients

DETAILED DESCRIPTION:
The proposed synopsis aims to compare the effectiveness of Alexander Technique nd Feldenkrais Technique in alleviating non spicific neck pain. Both AT and FT are somatic education methods focusing on improving body awareness and movement patterns. The study will involve non - specificc neck pain paytients randomly assigned to either AT Or FT intervention groups Outcome measures will include pain intensity, posture, functional ability and quality of sleep. Data will be collected at baseline, post - interventrion and on follow up to assess the short term and long term effects. Statistical analysis will be conducted to determine differences in outcomes between the two groups. Understanding the comparitive effectiveness of AT and FT could provide valuable insights for healthcare professionals in choosing appropriate intervention for non - specific neck pain patients management.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients
* Patients who have compromised activity of daily living due to neck pain
* Patients with non - specific neck pain
* Patients aging from 20 to 25 years

Exclusion Criteria:

* Patients with diagnose dneck pathologysuch as cervical disc herniation and spondylosis etc.
* Patients who are unable to participate in any physical activity
* Patients with recent neck injury or trauma
* Patients with cognitive impairment

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 22 Male Patients and 22 Female patients
Enrollment: 44 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Northwick Park Neck Pain Questionnaire | 4 Months
  The Northwick Park Neck Pain Questionnaire (NPQ) measures the neck pain and the consequent patient disabilities.
REEDCO Posture Assessment and Sleep Quality Scale | 4 Months
  a standard posture assessment and graded in the coronal and sagittal views in head-to-foot sequences

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No